CLINICAL TRIAL: NCT06057909
Title: Neurodegeneration and Neuronal Fluctuations in Lewy Body Disease and Alzheimer Disease
Brief Title: A Study of Neurodegeneration and Neuronal Fluctuations in Lewy Body Disease and Alzheimer's Disease
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Shannon Y. Chiu, Principal Investigator, Mayo Clinic
Other Study IDs: 23-007061; K23AG073525 (NIH)
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Lewy Body Disease; Alzheimer Disease; Healthy
MeSH Terms: conditions — Lewy Body Disease; Alzheimer Disease | interventions — Magnetic Resonance Imaging; Electroencephalography; Electromyography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Lewy Body Disease Group: Subjects identified by their physician with a diagnosis of Lewy body disease will have a physical and neurological exam, MRI of brain, electroencephalography (EEG), and electromyography (EMG).
  Interventions: Diagnostic Test: Magnetic Resonance Imaging; Diagnostic Test: Electroencephalography; Diagnostic Test: Electromyography
- Alzheimer Disease Group: Subjects identified by their physician with a diagnosis of Alzheimer will have a physical and neurological exam, MRI of brain, electroencephalography (EEG), and electromyography (EMG).
  Interventions: Diagnostic Test: Magnetic Resonance Imaging; Diagnostic Test: Electroencephalography; Diagnostic Test: Electromyography
- Healthy Control Group: Subjects identified as a health individual will have a physical and neurological exam, MRI of brain, electroencephalography (EEG), and electromyography (EMG).
  Interventions: Diagnostic Test: Magnetic Resonance Imaging; Diagnostic Test: Electroencephalography; Diagnostic Test: Electromyography

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging — Test that looks at the structure of the brain.
  Other Names: MRI
Diagnostic Test: Electroencephalography — Non-invasive technique to measure brain waves
  Other Names: EEG
Diagnostic Test: Electromyography — Technique to evaluate muscle activity
  Other Names: EMG

SUMMARY:
The purpose of this research study is to investigate how the brain, memory, thinking, and motor behavior change both in individuals with movement and/or cognitive disorders, as well as healthy individuals. Researchers will look at measurements of memory, thinking, brain wave and muscle activity, daily functioning, and brain scans to learn more about brain disorders such as Alzheimer disease and Lewy body disease.

ELIGIBILITY:
Inclusion Criteria:

* Use English as their primary language.
* Be willing to undergo health and cognitive assessments, as well as brain MRI and EEG study.
* Will be encouraged to have an available study partner (also called a "co-participant") who is familiar with the participant's daily functioning.
* This study will be limited to healthy individuals, and patients who have a clinical diagnosis made by a board-certified neurologist of Lewy body disease or Alzheimer disease.
* All individuals must be capable of providing informed consent and complying with the trial procedures. Realizing the challenge of obtaining informed consent from cognitively impaired individuals, time is specifically scheduled to foster an informative, supportive interview with the participant and caregiver/legal guardian (typically a spouse or child according to Arizona law and IRB guidelines).
* Ongoing participation will be maintained by strict adherence to inclusion/exclusion criteria, clinical appropriateness (as determined by participant's physician and proxy/family), as well as by expressed wishes of family members/caregivers/proxy discussed at each study visit (as appropriate).
* All participants will receive copies of the signed ICFs (including signatures of those obtaining consent).
* All participants have the right to withdraw from the study at any time.

Exclusion Criteria:

* Individuals will be excluded if they have significant sensory (visual and hearing) deficits or major medical or psychiatric illnesses which would limit participation.
* Participants will also be excluded if they have history of other major neurologic disorders including stroke, epilepsy, meningitis/encephalitis, metabolic or toxic encephalopathy, penetrating or severe closed head injury, brain tumor/other structural lesion, other primary movement disorders (such as essential tremor, dystonia, chorea, multiple system atrophy, progressive supranuclear palsy, corticobasal syndrome).
* In addition, as necessitated by the risks of Magnetic Resonance Imaging (MRI), patients who have any type of implanted electrical device (such as a cardiac pacemaker or a neurostimulator including deep brain stimulation), or a certain type of metallic clip in their body (i.e., an aneurysm clip in the brain), are not eligible for participation in the MRI portion of the study. Individuals who experience claustrophobic anxiety will also be excluded from participation.
* Women who are or might be pregnant and nursing mothers are not eligible.
* If the subject is a woman of childbearing potential, due to unknown risks to the fetus, they must have a pregnancy test. Individuals who have a history metalworking involving cutting processes such as grinding, filing, shaving, and threading, or history of eye injury involving metal, will also be excluded unless they have had prior documented radiological clearance for MRI.

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will include healthy individuals, and patients who have a clinical diagnosis made by a board-certified neurologist of Lewy body disease or Alzheimer disease.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Diffusion-weighted MRI (dMRI) | Baseline
  Measures diffusion of water molecules and cellular-level constraints
Electroencephalography (EEG) | Baseline
  Measures brain-wave activity

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Chiu, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials